CLINICAL TRIAL: NCT05712005
Title: Cognitive Testing in Diverse Populations to Further the Objective and Clinical Understanding of Cognivue Study (FOCUS)
Brief Title: Cognitive Testing in Diverse Populations to Further the Objective and Clinical Understanding of Cognivue Study
Acronym: FOCUS
Status: Completed | Type: Observational
Sponsor: Cognivue, Inc. (Industry)
Collaborators: Velocity Clinical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: COG-FOCUS
Record Dates: First submitted 2022-07-14; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Change
Keywords: cognition; brain neurology; neuropsychology; brain health; digital cognitive testing; digital biomarkers; computerized cognititve testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Study participants assigned to this group will complete the Cognivue 5-Minute Screening test across three domains including Memory, Visuospatial and Executive Function as well as two performance measures of Reaction Time and Speed Processing along with Normative Ranges 3 times OR study participants assigned to this group will complete the Cognivue 10-Minute Assessment test across six domains including Memory, Visuospatial, Executive Function, Naming/Language, Memory, Delayed Recall and Abstraction, as well as two performance measures of Reaction Time and Speed Processing, along with Normative Ranges 3 times. Next, study subjects will complete up to eight additional neuropsychological assessments, intermittently separated followed by the Cognivue Plus test.
- Group 2: Study subjects will complete up to eight additional neuropsychological assessments, intermittently separated followed by the Cognivue Plus test. Next, study participants assigned to this group will complete the Cognivue 5-Minute Screening test across three domains including Memory, Visuospatial and Executive Function as well as two performance measures of Reaction Time and Speed Processing along with Normative Ranges 3 times OR study participants assigned to this group will complete the Cognivue 10-Minute Assessment test across six domains including Memory, Visuospatial, Executive Function, Naming/Language, Memory, Delayed Recall and Abstraction, as well as two performance measures of Reaction Time and Speed Processing, along with Normative Ranges 3 times.
- Group 3: Study subjects will complete the Cognivue Plus test followed by completing up to eight additional neuropsychological assessments, intermittently separated. Next, study participants assigned to this group will complete the Cognivue 5-Minute Screening test across three domains including Memory, Visuospatial and Executive Function as well as two performance measures of Reaction Time and Speed Processing along with Normative Ranges 3 times OR study participants assigned to this group will complete the Cognivue 10-Minute Assessment test across six domains including Memory, Visuospatial, Executive Function, Naming/Language, Memory, Delayed Recall and Abstraction, as well as two performance measures of Reaction Time and Speed Processing, along with Normative Ranges 3 times.

SUMMARY:
An open-label, multi-site, validity and reliability study to obtain data on the Cognivue 5-Minute Screening and Cognivue 10-Minute Assessment tests to assess scoring and normative ranges and compare against other cognitive tests within a diverse population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Fluent in English
* Full vision in at least one eye
* Full use of at least one functional hand
* In overall good health, not experiencing any acute symptoms
* Agrees to cognitive examinations administered by research team

Exclusion Criteria:

* Age under 18
* Not fluent in English
* Blind in both eyes (any level of diagnosed blindness)
* Lacking a functional hand
* Those entering or in hospice
* Inability to agree to cognitive examinations administered by research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll up to 2,000 subjects at up to 20 study sites throughout the United States. Subjects will be divided into 6 age groups (i.e., 18-29; 30-39; 40-49; 50-59; 60-69; 70 and above). Subjects will complete one visit lasting up to two hours.
Sampling Method: Non-Probability Sample
Enrollment: 1437 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Confirmation of scoring and normative ranges. | 4 months
  Confirmation of scoring and normative ranges in Cognivue 5-Minute Screening and Cognivue 10-Minute Assessment tests.

SECONDARY OUTCOMES:
Stratify study population by age | 4 months
  Stratify study population by age compared to normative ranges of Cognivue 5-Minute Screening and Cognivue 10-Minute Assessment tests.
Stratify study population by sex | 4 months
  Stratify study population by sex compared to normative ranges of Cognivue 5-Minute Screening and Cognivue 10-Minute Assessment tests.
Stratify study population by education | 4 months
  Stratify study population by education compared to normative ranges of Cognivue 5-Minute Screening and Cognivue 10-Minute Assessment tests.
Stratify study population by ethnicity | 4 months
  Stratify study population by ethnicity compared to normative ranges of Cognivue 5-Minute Screening and Cognivue 10-Minute Assessment tests.
Training effect | 4 months
  Determine level of training effect.
Compare test sensitivity | 4 months
  Comparison of test sensitivity between Cognivue 5-Minute Screening and Cognivue 10-Minute Assessment tests and other cognitive assessment tests including: Reaction Time, Digit Span, Stroop and Visual Go No Go. In addition, RBANS and D-KEFS will be used as Cognitive Validators

CONTACTS AND LOCATIONS:
Overall Officials: James Galvin, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- Velocity Clinical Research, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.